CLINICAL TRIAL: NCT00000725
Title: A Phase I Study of AZT and Human Interferon Alpha (Recombinant Alpha-2A and Lymphoblastoid) in the Treatment of AIDS-Associated Kaposi's Sarcoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 013; 10989 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Sarcoma, Kaposi; HIV Infections
Keywords: Interferon Alfa-2a; Sarcoma, Kaposi; Dose-Response Relationship, Drug; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; Zidovudine; Interferon Type I
MeSH Terms: conditions — Sarcoma, Kaposi; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Interferon alpha-2; Zidovudine; interferon alfa-n1

INTERVENTIONS:
Drug: Interferon alfa-2a
Drug: Zidovudine
Drug: Interferon alfa-n1

SUMMARY:
To evaluate the safety and toxicity of combination therapy for AIDS-associated Kaposi's sarcoma with zidovudine (AZT) and two kinds of interferon alpha. The two kinds are interferon alpha (IFN-A) and interferon alpha-2A (recombinant) (IFN-A2A). To define the pharmacokinetics of both AZT and IFN-A or IFN-A2A when given in combination; to define the maximum tolerated dose of each drug in combination and to define doses to be used in Phase II trials. AZT has been found to inhibit both the in vitro (in test tube) and cell killing effects of HIV, and both interferons (IFN-A and IFN-A2A) have shown antiviral and antitumor effect in Kaposi's sarcoma. It is reasonable to assume that a synergistic effect and enhanced antitumor response may be seen with combination therapy. A study to evaluate the safety and efficacy of AZT in combination with IFN-A or IFN-A2A is warranted.

DETAILED DESCRIPTION:
AZT has been found to inhibit both the in vitro (in test tube) and cell killing effects of HIV, and both interferons (IFN-A and IFN-A2A) have shown antiviral and antitumor effect in Kaposi's sarcoma. It is reasonable to assume that a synergistic effect and enhanced antitumor response may be seen with combination therapy. A study to evaluate the safety and efficacy of AZT in combination with IFN-A or IFN-A2A is warranted.

Patients are randomized to receive IFN-A or IFN-A2A (given by intramuscular injection) and combined with AZT (taken orally) daily for 8 weeks. Study stops when maximum tolerated dose (MTD) is reached. Two cohorts of 4 patients enter each dose level. Patients do not enter into the next dose level until all patients have completed 3 weeks of treatment. AZT will escalate only if there is no unacceptable toxicity (grade 2 in = or > 3 patients or > grade 2 in any patient), subsequent increases in IFN-A or IFN-A2A will be permitted, but the AZT dose will remain fixed. The MTD for a given IFN-A or IFN-A2A dose level is defined as grade 2 toxicity (grade 3 for hemoglobin, neutrophil count, or SGOT) in 4 of the 6 patients. Patients have blood drawn every week and their general health is evaluated. Pharmacokinetic studies will be done on days 1, 21, and 24. Patients tolerating the combination may be continued on the same dose level for 1 year except if patient has reached complete remission for = or > 90 days, IFN-A or IFN-A2A will decrease to 3 times a week.

ELIGIBILITY:
Inclusion Criteria

* Patients must have biopsy-proven AIDS-associated Kaposi's sarcoma.
* Evidence of HIV infection as manifested by a positive antibody test.

Exclusion Criteria

* Active drug or alcohol abuse.

Co-existing Condition:

Excluded are patients with:

* Active opportunistic infections requiring ongoing therapy.
* Excluded within 90 days of study entry:
* Must be off therapy for Pneumocystis carinii pneumonia (PCP) unless recovered.
* Clinically significant cardiac disease, including a history of myocardial infarction or arrhythmia.
* Concurrent neoplasms other than basal cell carcinoma of the skin.
* Known hypersensitivity to polymycin B or neomycin.

Excluded are patients with:

* Active opportunistic infections requiring ongoing therapy.
* Excluded within 90 days of study entry:
* Must be off therapy for Pneumocystis carinii pneumonia (PCP) unless recovered.
* Clinically significant cardiac disease, including a history of myocardial infarction or arrhythmia.
* Concurrent neoplasms other than basal cell carcinoma of the skin.
* Known hypersensitivity to polymycin B or neomycin.

Prior Medication:

Excluded:

* Interferon.
* Zidovudine (AZT).
* Excluded within 30 days of study entry:
* Any biologic modifiers, corticosteroids, cytotoxic chemotherapeutic agents.
* Other drugs which can cause neutropenia or significant nephrotoxicity.
* Rifampin or rifampin derivatives, or systemic anti-infectives.
* Excluded within 90 days of study entry:
* Other antiviral agents.
* A history of Pneumocystis carinii pneumonia (PCP) completed treatment.

Prior Treatment:

Excluded within 30 days of study entry:

* Radiation therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56
Dates: Study Completion 1990-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fischl MA, Study Chair
Locations (1):
- Univ of Miami School of Medicine, Miami, Florida, United States

REFERENCES:
- [Background] Fischl MA, Uttamchandani RB, Resnick L, Agarwal R, Fletcher MA, Patrone-Reese J, Dearmas L, Chidekel J, McCann M, Myers M. A phase I study of recombinant human interferon-alpha 2a or human lymphoblastoid interferon-alpha n1 and concomitant zidovudine in patients with AIDS-related Kaposi's sarcoma. J Acquir Immune Defic Syndr (1988). 1991;4(1):1-10. PMID 1670585